CLINICAL TRIAL: NCT03047512
Title: Pilot Study of an Internet-based Program for Prevention and Early Intervention of Adolescent Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Henry Daniel Espinosa Duque, PhD, CES University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CES55384
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Depression
Keywords: Depression in adolescents; Mental Health; E-mental health; Prevention and Early intervention
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Pilot descriptive study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based program (Experimental): The internet based program includes the following modules: (1) information and psychoeducational material, (2) symptom monitoring with personalized automatic feedback, (3) forum (peer support moderated by mental health professionals) and (4) chat (individualized support by mental health professionals). It also considers (5) the referral to face-to-face treatment of cases with symptoms that require it. (6) In addition to the web page in the institutions, there will be a monthly health promotion booth during breaks.
  Interventions: Behavioral: Experimental: Internet-based program
- Control Group (No Intervention): The control group will receive two psychoeducational workshops / conferences. In addition, the adolescents in the control group can participate in the monthly health promotion booths offered by the program.

INTERVENTIONS:
Behavioral: Experimental: Internet-based program — * Adolescents who obtain a score between 2 and 4 on the PHQ-3 will be invited to use the information module, the psychoeducational material and the symptom monitoring with personalized automatic feedback.
  * Adolescents who obtain a score between 5 and 6 on the PHQ-3 will be invited to use, in addition to the above, group forum activities (peer support moderated by mental health professionals) and the possibility of a chat (individualized support by mental health professionals).
  * Adolescents who obtain a score greater than 6 on the PHQ-3 or that have suicidal thoughts will be invited to see the mental health counselor of the institution and the possibility of their reference to face-to-face professional attention will be considered.
  Other Names: Cuida tu Animo active group
  Arms: Internet-based program

SUMMARY:
Major depression is a highly prevalent and severe mental disease that negatively alters the lives of people, their families, and their social environment.

Organizations that promote mental health policies have recognized the potential of new information technologies for the prevention and treatment of mental disorders. In this direction, information and communication technologies (ICTs) generate opportunities for increasing patient well-being through the use of on-line software. Such programs often include interactivity, self-monitoring, information materials (sometimes in multimedia format), and exercises on problem solving, recognition and challenging of dysfunctional thoughts, scheduling of activities, behavioral experiments, and other psycho-educational activities.

In Colombia, there are few preventive mental health interventions scientifically oriented and seeking to demonstrate efficacy in context.

The purpose of this study is to determine whether an internet-based program is effective to prevent and to intervene early the depression in adolescents between 11 and 20 years of age in 2 schools in the Antioquia Region, Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who study in schools in Antioquia from sixth grade to tenth grade, who can access the internet and a psychological service in case of moderate or severe depressive symptoms.

Exclusion Criteria:

* High suicide risk defined by: A score equal to or greater than 2 in the question 9 of the PHQ-9A, an adolescent who is undergoing treatment with antidepressants and / or currently attends psychotherapy

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 213 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Depressive Symptomatology | Baseline, 4 months, 12 months
  Depressive symptomatology measured with the Patient Health Questionnaire PHQ -9

SECONDARY OUTCOMES:
Change from Baseline in Health Related Quality | Baseline, 4 months, 12 months
  Health Related Quality of Life Questionnaire for Children and Young People KIDSCREEN-10
Change from Baseline in anxious symptoms | Baseline, 4 months, 12 months
  Generalised Anxiety Disorder Assessment (GAD-7)
Change from Baseline in of depression | Baseline, 4 months, 12 month
  Self-Stigma of Depression Scale (SSDS)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Espinosa, PhD, Study Director — CES University
Locations (8):
- Colombia (8):
  - Institucion Educativa El Perpetuo Socorro, Medellín, Antioquia
  - Institucion Educativa El Salvador, Medellín, Antioquia
  - Institución Educativa America, Medellín, Antioquia
  - Institución Educativa El Corazón, Medellín, Antioquia
  - Institución Educativa Fatima Nutibara, Medellín, Antioquia
  - Institución Educativa Francisco Antonio Zea, Medellín, Antioquia
  - Institución Educativa Mariscal Robledo, Medellín, Antioquia
  - Institución Educativa Villa Flora, Medellín, Antioquia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sobocki P, Jonsson B, Angst J, Rehnberg C. Cost of depression in Europe. J Ment Health Policy Econ. 2006 Jun;9(2):87-98. PMID 17007486
- [Background] Vargas-Zea N, Castro H, Rodriguez-Paez F, Tellez D, Salazar-Arias R. Colombian Health System on its Way to Improve Allocation Efficiency-Transition from a Health Sector Reform to the Settlement of an HTA Agency. Value Health Reg Issues. 2012 Dec;1(2):218-222. doi: 10.1016/j.vhri.2012.09.004. Epub 2012 Dec 12. PMID 29702903
- [Background] Barney LJ, Griffiths KM, Christensen H, Jorm AF. The Self-Stigma of Depression Scale (SSDS): development and psychometric evaluation of a new instrument. Int J Methods Psychiatr Res. 2010 Dec;19(4):243-54. doi: 10.1002/mpr.325. PMID 20683846
- [Background] Fernández, J. & Gómez-Restrepo, C. Telepsiquiatría: innovación de la atención en salud mental. Una perspectiva general. Rev. Colomb. Psiquiat., 40 (3), 2011.
- [Background] Collins PY, Patel V, Joestl SS, March D, Insel TR, Daar AS; Scientific Advisory Board and the Executive Committee of the Grand Challenges on Global Mental Health; Anderson W, Dhansay MA, Phillips A, Shurin S, Walport M, Ewart W, Savill SJ, Bordin IA, Costello EJ, Durkin M, Fairburn C, Glass RI, Hall W, Huang Y, Hyman SE, Jamison K, Kaaya S, Kapur S, Kleinman A, Ogunniyi A, Otero-Ojeda A, Poo MM, Ravindranath V, Sahakian BJ, Saxena S, Singer PA, Stein DJ. Grand challenges in global mental health. Nature. 2011 Jul 6;475(7354):27-30. doi: 10.1038/475027a. No abstract available. PMID 21734685
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Moras, K. Twenty-five years of psychological treatment research on unipolar depression in adult outpatients: Introduction to the special section. Psychotherapy Research , 16 (5), 519-525, 2006.
- [Background] Proudfoot JG. Computer-based treatment for anxiety and depression: is it feasible? Is it effective? Neurosci Biobehav Rev. 2004 May;28(3):353-63. doi: 10.1016/j.neubiorev.2004.03.008. PMID 15225977
- [Background] Richardson LP, McCauley E, Grossman DC, McCarty CA, Richards J, Russo JE, Rockhill C, Katon W. Evaluation of the Patient Health Questionnaire-9 Item for detecting major depression among adolescents. Pediatrics. 2010 Dec;126(6):1117-23. doi: 10.1542/peds.2010-0852. Epub 2010 Nov 1. PMID 21041282
- [Background] KIDSCREEN Group Europe. The KIDSCREEN questionnaires. Quality of life questionnaires for children and adolescents- Handbook. Lengerich, Germany: Papst Science Publisher. 2006.